CLINICAL TRIAL: NCT06110000
Title: Effects of Pragmatic Set of Interventions Versus Scapular Strengthening Exercises on Scapular Dyskinesia in Adhesive Capsulitis
Brief Title: Pragmatic Set of Interventions Versus Scapular Strengthening Exercises on Scapular Dyskinesia in Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0150
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Scapular Dyskinesis; Adhesive Capsulitis
Keywords: Scapular Dyskinesis; Adhesive Capsulitis; Pragmatic set of interventions; strengthening exercise
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Participants are divided into two groups. Group A assigned to pragmatic group of interventions and group B assigned with scapular strengthening exercises at the beginning of the trial and continue that throughout the length of the trial.
Who Masked: Participant
Masking Description: Blinding,refers to a practice where study participants are prevented from knowing certain information that may somehow influence them-thereby tainting the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pragmatic set of interventions (Experimental): The pragmatic set included 6 interventions as follows.
  1. Pragmatic posterior capsular stretch (PPCS)
  2. Serratus anterior stretch (SAS)
  3. Rotator cuff facilitation (RCF)
  4. Acromioclavicular joint mobilization
  5. Pectoralis minor stretch
  6. Thoracic manipulation
  Interventions: Other: pragmatic set of interventipons
- scapular strengthening exercises (Placebo Comparator): Scapular strengthening exercises will be individualised focusing on Serratus anterior, trapezius, Levator scapulae, Rhomboids.
  Serratus anterior;
  * Dynamic hug
  * Scaption with external rotation
  * Diagonal PNF (shoulder flexion, horizontal flexion, external rotation),
  Trapezius - Upper trapezius:
  * Unilateral shoulder shrug,
  * Rowing,
  * Forward shoulder flexion,
  * Shoulder abduction in scapular plane above 120 degrees.
  Middle trapezius:
  * Prone shoulder horizontal abduction
  * Scaption, horizontal abduction with external rotation
  Lower trapezius:
  * Unilateral scapular retraction,
  * Prone bilateral shoulder external rotation at 90 degrees of abduction,
  * Prone shoulder abduction.
  Levator Scapulae:
  * Horizontal abduction with shrug,
  * Horizontal abduction with ER,
  * Prone shoulder extension.
  Rhomboids:
  * ER at 90° of abduction,
  * ER at 0° of abduction,
  * Horizontal abduction,
  * Shoulder extension,
  Interventions: Other: scapular strengthening exercise.

INTERVENTIONS:
Other: pragmatic set of interventipons — The pragmatic set included 6 interventions as follows.
  1. Pragmatic posterior capsular stretch (PPCS)
  2. Serratus anterior stretch (SAS)
  3. Rotator cuff facilitation (RCF)
  4. Acromioclavicular joint mobilization.
  5. Pectoralis minor stretch
  6. Thoracic manipulation Five to ten sweeps per minute are administered three to four times. The applied force is combined with deep breathing. The subject is asked to report discomfort and the applied force is adjusted.
  Arms: pragmatic set of interventions
Other: scapular strengthening exercise. — • Subjects in Group B receive strengthening exercises (exercise will perform with 15 repetitions for each set- 3sets/day, 3 days /week for 6 weeks. In Scapular strengthening exercises, treatment protocol will involve the individualized for focus muscle Serratus anterior (Dynamic hug, Scaption with external rotation, Diagonal PNF (shoulder flexion horizontal flexion, external rotation),Trapezius - Upper trapezius (unilateral shoulder shrug, rowing, forward shoulder flexion, shoulder abduction in scapular plane above 120 degrees, Middle trapezius (prone shoulder horizontal abduction, scaption, horizontal abduction with external rotation), Lower trapezius (Unilateral scapular retraction, prone bilateral shoulder external rotation at 90 degrees of abduction, prone shoulder abduction), Levator Scapulae (horizontal abduction with shrug, horizontal abduction with ER, prone shoulder extension, Rhomboids (ER at 90° of abduction, ER at 0° of abduction, Horizontal abduction, Shoulder extension)
  Arms: scapular strengthening exercises

SUMMARY:
The aim of this study is to determine the Effects of pragmatic set of interventions versus scapular strengthening exercises on scapular dyskinesia in adhesive capsulitis.

DETAILED DESCRIPTION:
Scapular dyskinesia (SD) is a term that describes a physical impairment in which the scapula's position and motion are altered.Symptoms of SD can be one or a combination of the anterior shoulder pain, Postero-superior scapular pain, superior shoulder pain, proximal lateral arm pain. scapular dyskinesia is commonly found in adhesive capsulitis patients. To determine the scapular dyskinesia with shoulder pain two tests that apply manual assistance to the scapula are lateral scapular slide test and wall push up test.

Pragmatic set of interventions are an important element in rehabilitation, and has improved the treatment of many musculoskeletal and neurological conditions. Scapular strengthening exercises, which aims to improve abnormal scapular movements that commonly occur in people with adhesive capsulitis.

The purpose of this study is to explore the effect of scapular focused exercises on the rehabilitation of adhesive capsulitis, patient with scapular dyskinesia. The importance of scapular rehabilitation in the treatment of scapular dyskinesia and to examine the comparative effect of pragmatic set of intervention with scapular strengthening protocol on scapular dyskinesia.

My study on the effect of a pragmatic set of intervention versus scapular strengthening exercises on scapular dyskinesia in adhesive capsulitis is important because it addresses a gap in the current literature. While both interventions have been shown to improve scapular dyskinesia in patients with adhesive capsulitis, there is a lack of studies comparing the two methods. My study will help determine which intervention is more effective in treating scapular dyskinesia, which will be valuable information for healthcare providers working with patients with adhesive capsulitis

ELIGIBILITY:
Inclusion Criteria:

* Both male and females with age range b/w 25-45
* People with adhesive capsulitis (having pain, stiffness, and decrease movements of - external rotation, forward flexion and abduction)
* Scapular dyskinesia (positive lateral scapular slide with difference of 1.5cm when measurements are compared bilaterally)

Exclusion Criteria:

* History of shoulder surgery or other significant shoulder injury, neurological or musculoskeletal conditions that may affect shoulder function.
* History of significant medical conditions (e.g., heart disease, cancer) that may affect their ability to participate in the study.
* Pregnant or breast feeder, as the exercise program may not be safe or appropriate for them.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | 4th week
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. SPADI was found to have reliability coefficients of ICC ≥ 0.89 in a variety of patient populations.Internal consistency is high with Cronbach α typically exceeding 0.90. The SPADI demonstrates good construct validity, correlating well with other region-specific shoulder questionnaires.
Scapulometer | 4th week
  is a reliable tool to measure scapular medial border and inferior angle prominence. It is used to measure the distance from the root of the spine (ROS) and the inferior angle (INF) of the scapula to the thorax wall. The novel scapulometer has excellent reliability and fair validity to quantify medial border and inferior angle prominence of the scapula. Further research utilizing this instrument is recommended.

SECONDARY OUTCOMES:
Visual analogue scale: | 4th week
  This VAS will be used in this study to measure Pain. Patients were instructed to assess the severity of shoulder pain experienced last week on a 0-10 cm horizontal line (0 = painless and 10 = worst pain imaginable). The VAS has been shown to have excellent test-retest reliability (ICC = 0.97) and high validity (r with a 5-point verbal descriptive scale = 0.71-0.78) to evaluate pain perception.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, Phd, Principal Investigator — Riphah International University
Locations (1):
- Amina welfare and Trust, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Background] Mohamed AA, Alawna M. Effect of Adding Vertical Correction to Dynamic Scapular Recognition on Scapular Dyskinesis and Shoulder Disability in Patients With Adhesive Capsulitis: A Randomized Clinical Study. J Chiropr Med. 2022 Jun;21(2):124-135. doi: 10.1016/j.jcm.2022.02.002. Epub 2022 Apr 4. PMID 35774629
- [Background] Zhu Y, Blundell JE, Holschuh NM, McLean R, Menon RS. Validation of a Mobile App-Based Visual Analog Scale for Appetite Measurement in the Real World: A Randomized Digital Clinical Trial. Nutrients. 2023 Jan 7;15(2):304. doi: 10.3390/nu15020304. PMID 36678176
- [Background] Lluch-Girbes E, Requejo-Salinas N, Fernandez-Matias R, Revert E, Vila Mejias M, Rezende Camargo P, Jaggi A, Sciascia A, Horsley I, Pontillo M, Gibson J, Richardson E, Johansson F, Maenhout A, Oliver GD, Turgut E, Jayaraman C, Duzgun I, Borms D, Ellenbecker T, Cools A. Kinetic chain revisited: consensus expert opinion on terminology, clinical reasoning, examination, and treatment in people with shoulder pain. J Shoulder Elbow Surg. 2023 Aug;32(8):e415-e428. doi: 10.1016/j.jse.2023.01.018. Epub 2023 Feb 15. PMID 36796714
- [Background] Dube MO, Desmeules F, Lewis JS, Roy JS. Does the addition of motor control or strengthening exercises to education result in better outcomes for rotator cuff-related shoulder pain? A multiarm randomised controlled trial. Br J Sports Med. 2023 Apr;57(8):457-463. doi: 10.1136/bjsports-2021-105027. Epub 2023 Feb 16. PMID 36796859
- [Background] Karaagac A, Arslan SA, Keskin ED. Assessment of pain, scapulothoracic muscle strength, endurance and scapular dyskinesis in individuals with and without nonspecific chronic neck pain: A cross-sectional study. J Bodyw Mov Ther. 2023 Jul;35:261-267. doi: 10.1016/j.jbmt.2023.04.008. Epub 2023 Apr 19. PMID 37330779
- [Background] Ucurum SG, Karabay D, Ozturk BB, Kaya DO. Comparison of scapular position and upper extremity muscle strength in patients with and without lateral epicondylalgia: a case-control study. J Shoulder Elbow Surg. 2019 Jun;28(6):1111-1119. doi: 10.1016/j.jse.2018.12.010. Epub 2019 Mar 26. PMID 30926184